CLINICAL TRIAL: NCT04466553
Title: MIS Hematoma Evacuation
Status: Withdrawn | Type: Observational
Why Stopped: The study did not begin.
Sponsor: Lahey Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 20203097
Record Dates: First submitted 2020-07-01; First posted 2020-07-10 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Intracranial Hematoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- NICO BrainPath™ Patients: 50 patients will be enrolled in Group A NICO BrainPath™ system.
  The NICO BrainPath™ System has been proposed to reduce high morbidity and mortality associated with ICH through minimally invasive clot evacuation. Previous, single-center trials concluded evacuation of ICH using the BrainPath™ system as being safe and effective. Additionally, previous studies concluded that lesser ICH removal was correlated with mortality benefit and that the NICO BrainPath™ system approach was shown to be safe and effective with a high rate of clot evacuation and functional independence. This system warrants further research because of the need to optimize clinical outcome in these patients and to better define the role of hematoma evacuation in the care of these patients.
  Interventions: Device: NICO BrainPath™ System
- Standard of Care: 50 patients will be matched retrospectively of similar diagnosis, undergoing standard of care (e.g. no surgical intervention). These patients will be matched to the surgical patients based on age, gender, and location of hemorrhage.

INTERVENTIONS:
Device: NICO BrainPath™ System — Patients who are admitted under the neurology service in the Neurocritical Care and Medical ICU will be screened for participation in the trial by their treating physician. Once blood pressure has been stabilized and the best medical treatment has been determined, the patient will need to undergo a standard of care, repeat CT scan 6 hours after stabilization to show that there has been no increase in size of the ICH. Patients that meet eligibility criteria after this CT will be taken to the OR within 24-72 hours for a minimally invasive, navigation guided endoport based evacuation of the clot using the NICO BrainPath™ system.
  Groups: NICO BrainPath™ Patients

SUMMARY:
The primary objective of this study is to determine the effectiveness of the NICO BrainPath™ hematoma evacuation system for patients between the ages of 18 and 80 years old with an intracerebral hematoma. Effectiveness will be defined as the ability to achieve either 70% reduction of intracranial hematoma or to achieve <15 ml residual hematoma volume following surgery.

Additionally, the study aims to compare the mortality and complication rate of patients who undergo minimally invasive, navigation guided endoport based evacuation of intracerebral hematoma with NICO BrainPath™ System as compared to non-operative, supportive standard of care.

The study is a prospective, non-randomized cohort study. 50 patients will be enrolled in Group A (NICO BrainPath™ system) and 50 patients will be matched retrospectively of similar diagnosis, undergoing standard of care from Epic). 50 patients will undergo minimally invasive, navigation guided endport based evacuation of intracerebral hematoma with NICO BrainPath™ System. The patient population receiving non-operative supportive care will be matched to the surgical patients based on age, gender, and location of hemorrhage.

DETAILED DESCRIPTION:
Approximately 100 patients will participate in this study. Patients with significant intraparenchymal hemorrhage who are admitted under the neurology service in the Neurocritical Care and Medical ICU will be screened for eligibility.

A repeat CT scan 6 hours after stabilization to show that there has been no increase in size of the ICH will determine eligibility in the trial. Patients that meet eligibility criteria after this CT will be taken to the OR within 24-72 hours for a minimally invasive, navigation guided endoport based evacuation of the clot using the NICO BrainPath™ system.

At baseline, the Glasgow Coma Scale (GCS) and the Modified Rankin Score (mRS) will be captured, along with baseline demographics. The GCS and mRS will be recorded at 1-, 3, and 6-month post-operatively. A follow-up CT will be captured at 3 months. Mortality and adverse events will be reviewed at each timepoint.

ELIGIBILITY:
Inclusion Criteria:

1. 18 and 80 years of age, inclusive
2. Spontaneous supratentorial, intracerebral hematoma ICH >30 ml measured by the ABC/2 method.
3. Location of Hemorrhage: Lobar, Putaminal and/or Caudate
4. A Glasgow Coma Scale (GCS) of 4 or greater
5. Historical Modified Rankin Score (mRS) of 0 (no symptoms of neurological disability) or 1 (no significant disability despite symptoms, able to carry out usual duties and activities).

Exclusion Criteria:

1. Pupils dilated and fixed
2. Rapidly deteriorating patient (at the discretion of the surgeon)
3. Primary Thalamic Bleed
4. Intraventricular Blood (more than 50 % of either ventricle, visual estimate)
5. ICH secondary to aneurysm
6. Arteriovenous malformation (AVM)
7. Tumor
8. Moya-Moya
9. Sinus thrombosis
10. Platelet count <100,000, INR >1.4
11. Known coagulopathy, on anticoagulants that cannot be reversed

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Male and females between the ages of 18-80 years old.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of the NICO BrainPath™ hematoma evacuation system | immediately after the surgery.
  The primary objective of this study is to determine the effectiveness of the NICO BrainPath™ hematoma evacuation system for patients between the ages of 18 and 80 years old with an intracerebral hematoma. Effectiveness will be defined as the ability to achieve either 70% reduction of intracranial hematoma or to achieve <15 ml residual hematoma volume immediately after the surgery.

SECONDARY OUTCOMES:
Comparison of mortality and complication rate. | 6 months post-op
  Additionally, the study aims to compare the mortality and complication rate of patients who undergo minimally invasive, navigation guided endoport based evacuation of intracerebral hematoma with NICO BrainPath™ System as compared to non-operative, supportive standard of care until six months post-operative.

CONTACTS AND LOCATIONS:
Overall Officials: Haran Ramachandran, MD, Principal Investigator — Lahey Clinic; Zoher Ghogawala, MD, Study Chair — Lahey Clinic

IPD SHARING:
Plan to Share IPD: Undecided